CLINICAL TRIAL: NCT02431117
Title: A Multicenter, Longitudinal, Non-drug Study to Assess the Suitability of Neurocognitive Tests and Functioning Scales for the Measurement of Cognitive and Functioning Changes in Japanese Individuals With Down Syndrome Aged 6-30
Brief Title: Non-drug Study to Assess the Suitability of Assessment Scales in Japanese Individuals With Down Syndrome Aged 6-30
Status: Completed | Type: Observational
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: JP29688
Record Dates: First submitted 2015-04-13; First posted 2015-04-30 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To evaluate the suitability (i.e. number of tests completed and number of participants completing the tests, variance estimate of baseline and of the change from baseline values) of neurocognitive tests and functioning scales in view of their use in future multicenter, multinational clinical efficacy trials testing a putative cognitive enhancer for individuals with Down syndrome aged 6-30.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may have standard trisomy 21, Robertsonian translocation, isochromosome21,Down syndrome with reciprocal translocation or mosaicism.
* Availability of parent or other reliable caregiver who agrees to accompany the subject to clinic visits, provide information about the subject's behavior and symptoms.
* Down Syndrome subjects meeting clinical diagnostic criteria for generalized anxiety disorders, major depressive disorders, autism spectrum disorder, attention deficit and hyperactivity disorder, can participate to the study provided they are on stable medication for at least 8 weeks prior to screening.

Exclusion Criteria:

Individuals who may not be able to comply with the protocol or perform the outcome measures due to significant hearing or visual impairment or other issues judged relevant by the investigators.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: People with Down syndrome
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Suitability for individuals with Down syndrome assessed by number of tests completed and number of participants completing the tests, variance estimate of baseline and of the change from baseline values. | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hideaki Takahashi, Study Director — Chugai Pharmaceutical
Locations (7):
- Japan (7):
  - Sapporo, Hokkaido
  - Yokohama, Kanagawa
  - Izumi, Osaka
  - Takatsuki, Osaka
  - Saitama, Saitama
  - Chiyoda-ku, Tokyo
  - Setagaya-ku, Tokyo